CLINICAL TRIAL: NCT05507840
Title: Photobiomodulation for Dry Age Related Macula Degeneration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, ANCA ROALD, Principal Investigator, MD dr. med., Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 456056
Record Dates: First submitted 2022-06-30; First posted 2022-08-19 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Photobiomodulation; Age-Related Macular Degeneration
Keywords: choroidal neovascular membrane
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Near or infra red light provided by the Valeda machine will be applied in the intervention eye
  Interventions: Device: Valeda machine
- Control (Sham Comparator): Light with very low intensity provided by the same Valeda machine will be applied in the control eye
  Interventions: Device: Valeda machine

INTERVENTIONS:
Device: Valeda machine — Photobiomodulation treatment with Valeda machine will be applied every six months for 2 years in patients with dry age related macula degeneration.

SUMMARY:
The study will investigate the effect of photobiomodulation treatment on the risk of developing late age related macula degeneration (AMD) in the study eye in patients with wet AMD in the fellow eye.

ELIGIBILITY:
Inclusion Criteria:

* patients with dry AMD in the study eye and wet AMD in the control eye

Exclusion Criteria:

* Geographic atrophy of the central macular region at enrolment
* Previous/ active wet AMD in the study eye
* A history of epilepsy
* Retinal diseases apart from AMD
* Significant media opacities
* Cataracts worse than grade 2 (LOCS III classification)
* Change in AREDS 2 supplements (vitamins) 1 month before the study and during the study trial was allowed.
* Ongoing systemic medications that are photosensitizing (e.g. tetracyclins)
* Systemic medications during the last 6 months that can cause deposits in the macular region (hydroxychloroquine, amiodarone)
* Unable to give informed consent
* Unable to cooperate with the treatment and follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that develope late AMD in the study eye compared with control after 3 years of follow-up | 3 years